CLINICAL TRIAL: NCT01496755
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled Trial of Single and Multiple Doses of RG7667 in Healthy Adult Volunteers
Brief Title: A Study of RG7667 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GV28012
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — RG7667

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RG7667 (Experimental)
  Interventions: Drug: RG7667

INTERVENTIONS:
Drug: Placebo — Single/multiple doses
  Arms: Placebo
Drug: RG7667 — Single/multiple ascending doses
  Arms: RG7667

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the safety and pharmacokinetics of RG7667 in healthy volunteers. Subjects will be randomized in cohorts to receive either single/multiple doses of RG7667 intravenously or placebo. Anticipated time on study treatment is up to 57 days with a 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 to 55 years of age, inclusive
* Body mass index 18.0 to 31.0 kg/m2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, vital signs, and laboratory values, as deemed by the Investigator

Exclusion Criteria:

* History of malignancy, except completely excised basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ
* History of severe bacterial, fungal, or parasitic infections (more than 2 hospitalizations within 1 year or more than 2 courses of iv antibiotics within 1 year)
* Pregnant, lactating, or planned pregnancy within 6 months of Screening
* Positive for hepatitis B, hepatitis C or HIV infection
* Exposure to any investigational biological agent within 90 days prior to the Screening evaluation or received any other investigational treatment 30 days prior to the Screening evaluation (or within 5 half-lives of the investigational agent, whichever is greater)
* History of alcoholism or drug addiction within 1 year of Screening
* Positive urine test for selected drugs of abuse at Screening and Check-in (Day -1); positive breathalyzer test for alcohol at Check-in
* Use of prescription drugs within 14 days prior to Day 1 or during the study, except for hormonal contraceptives or hormone replacement therapy
* Use of over-the-counter (OTC) medication within 7 days prior to Day 1 or during the study. Medications such as acetaminophen and ibuprofen and routinely-taken dietary supplements, including vitamins and herbal supplements are allowed at the discretion of the investigator and Sponsor.
* Donation of plasma within 7 days prior to Day 1. Donation or loss of blood of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to Day 1.
* Lack of peripheral venous access

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to 141 days

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | up to 141 days
Pharmacokinetic: Maximum serum concentration (Cmax) | up to 141 days
Pharmacokinetic: Time to maximum serum concentration (tmax) | up to 141 days
Pharmacokinetic: Apparent clearance (CL/F) | up to 141 days
Pharmacokinetic: Terminal half-life (t½) | up to 141 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - Daytona Beach, Florida
  - Honolulu, Hawaii
  - Evansville, Indiana
  - Dallas, Texas
  - Madison, Wisconsin

REFERENCES:
- [Derived] Ishida JH, Burgess T, Derby MA, Brown PA, Maia M, Deng R, Emu B, Feierbach B, Fouts AE, Liao XC, Tavel JA. Phase 1 Randomized, Double-Blind, Placebo-Controlled Study of RG7667, an Anticytomegalovirus Combination Monoclonal Antibody Therapy, in Healthy Adults. Antimicrob Agents Chemother. 2015 Aug;59(8):4919-29. doi: 10.1128/AAC.00523-15. Epub 2015 Jun 8. PMID 26055360